CLINICAL TRIAL: NCT02102880
Title: The Role of Complement Factor H Polymorphism in the Regulation of Choroidal Vascular Tone in Young Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Ass.Prof.Dr.med., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPHT-040214
Record Dates: First submitted 2014-03-21; First posted 2014-04-03 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Age-Related Macular Degeneration
Keywords: Genetic Association Studies
MeSH Terms: conditions — Macular Degeneration

ARMS (1):
- Healthy Subjects (Other)
  Interventions: Genetic: the polymerase chain reaction (PCR)

INTERVENTIONS:
Genetic: the polymerase chain reaction (PCR)

SUMMARY:
Age related macular degeneration (AMD) is a multifactorial disease with a strong genetic component. Given that it is known that impaired regulation of choroidal vascular tone is present in patients with AMD, the current study seeks to investigate whether genetic polymorphisms in risk alleles for AMD are associated with altered choroidal blood flow regulation in healthy subjects. For this purpose a total of 220 healthy volunteers will be included. Choroidal blood flow regulation will be evaluated by measuring choroidal blood flow during isometric exercise. In addition, flicker induced vasodilatation will be studied and retinal vessel calibers will assessed, as well as retinal thickness and macular pigment optical density.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 45 years, nonsmokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Systolic blood pressure < 160 mmHg, diastolic blood pressure < 90 mmHg
* Normal ophthalmic findings, ametropia less than 3 diopters

Exclusion Criteria:

* Regular use of medication
* Abuse of alcoholic beverages
* Participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except hormonal contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* History or family history of epilepsy
* Pregnancy, planned pregnancy or lactating

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2023-09-02 (Estimated); Study Completion 2023-09-02 (Estimated)

PRIMARY OUTCOMES:
Choroidal blood flow during isometric exercise (LDF) | 1 day

SECONDARY OUTCOMES:
Flicker induced vasodilatation, expressed as percent change to baseline (DVA) | 1 day
Genotyping (PCR) | 1 day
Retinal vessel calibers and AV- ratio (DVA) | 1 day
Laser Speckle Flowmetry (LSFG) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Calzetti G, Fondi K, Bata AM, Luft N, Wozniak PA, Witkowska KJ, Bolz M, Popa-Cherecheanu A, Werkmeister RM, Schmidl D, Garhofer G, Schmetterer L. Assessment of choroidal blood flow using laser speckle flowgraphy. Br J Ophthalmol. 2018 Dec;102(12):1679-1683. doi: 10.1136/bjophthalmol-2017-311750. Epub 2018 Feb 22. PMID 29472236
- [Derived] Witkowska KJ, Bata AM, Calzetti G, Luft N, Fondi K, Wozniak PA, Schmidl D, Bolz M, Popa-Cherecheanu A, Werkmeister RM, Garhofer G, Schmetterer L. Optic nerve head and retinal blood flow regulation during isometric exercise as assessed with laser speckle flowgraphy. PLoS One. 2017 Sep 12;12(9):e0184772. doi: 10.1371/journal.pone.0184772. eCollection 2017. PMID 28898284